CLINICAL TRIAL: NCT04975841
Title: Inclusion Body Myositis Treatment With Celution Processed Adipose Derived Regenerative Cells
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: IBM-ADRC
Record Dates: First submitted 2020-11-09; First posted 2021-07-23 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Inclusion Body Myositis
Keywords: IBM
MeSH Terms: conditions — Myositis, Inclusion Body

STUDY DESIGN:
Intervention Model Description: Six subjects will be randomized to Part 1 and start Part 2 once Part 1 is completed. Three subjects will be randomized directly to Part 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Standard of Care (No Intervention): Standard of Care (SOC) Study: The 6 subjects in the late injection group will start on Part 1. - The Part 1 study subject participation is 12 months. Two subjects will be enrolled at each of Months 0, 3 and 6. This will include an initial assessment and SOC follow-up. Subjects will continue standard of care treatment. Part 1 study duration (with staggering included) will be 18 months. After Part 1, the late injection subjects may proceed to Part 2 depending on safety data from the early injection group (see 3. below).
- Stem Cell Injection (Active Comparator): Stem Cell Injection: The three subjects randomized to early injections will proceed directly to Part 2 with staggered enrollment of 1 subject every 3 months. Once the safety data of the first subject at Month 3 is assessed, the second subject will be enrolled. Once the safety data of the first 2 subject (Subject 1 at Month 6 and Subject 2 at Month 3) are assessed, the third early injection subject will be enrolled in Part 2.
  Interventions: Device: Adipose Derived Regenerative Cells

INTERVENTIONS:
Device: Adipose Derived Regenerative Cells — The Cytori Celution technology is an automated version of the process and techniques used in the research laboratory to isolate regenerative cells from adipose tissue. The Cytori Celution System uses a proteolytic enzyme blend (Celase) to disrupt the adipose tissue matrix and release the entrapped adipose derived regenerative cells (ADRCs), also referred to in the literature as "stromal vascular fraction" cells. Once digested, the digestate is separated into fractions (buoyant adipocytes (fat cells) and pelleted ADRCs) by centrifugation. The non-buoyant cell pellet (ADRCs) is then washed and centrifuged through several cycles to remove residual enzyme reagent and cellular debris. Although the Cytori Celution technology replicates known laboratory techniques, it offers significant improvements to the manual laboratory technique by controlling the processing in a closed system that has been validated for safety, performance, and reproducibility.
  Arms: Stem Cell Injection

SUMMARY:
This is an open-label, single arm study evaluating the safety for patients with Inclusion Body Myositis. A total of 9 subjects will be enrolled in the study. Subjects will be randomized to Part 1 or Part 2 of the study in blocks of 3 every 3 months. Stem cell injections will be given in the forearm and thigh on either the left or right side of the body, depending on which side meets criteria. The overall goal of this pilot study is to test the safety of adipose derived regenerative cells in patients with Inclusion Body Myositis. If determined safe, this trial could lead to larger Phase II trials. While this specific trial's primary endpoint is safety, it our ultimate hope that ADRC injections into the forearm and thigh of IBM patients will slow, stabilize, or even reverse the progression of muscle weakness in patients with IBM.

DETAILED DESCRIPTION:
Inclusion Body Myositis (IBM) is the most common progressive and debilitating muscle disease beginning in persons over age 50 years, with an annual incidence estimated at 2.2 to 7.9 per million. IBM causes both proximal and distal muscle weakness, characteristically most prominent in the quadriceps and finger flexors. Over time it can lead to severe disability, including loss of hand function, falls due to quadriceps muscle weakness and foot drop, dysphagia, and eventually respiratory muscle weakness. There is no effective therapy for IBM.

This study, "Inclusion Body Myositis Treatment with Celution Processed Adipose Derived Regenerative Cells" (IBM-ADRC) evaluates the safety and efficacy of the Celution System in the processing of an autologous graft consisting of adipose-derived regenerative cells (ADRCs) in the treatment of inclusion body myositis. Specifically, the overall objective is for the proposed clinical trial to serve as a safety trial for Inclusion Body Myositis.

This is an open-label, single arm study evaluating the safety for patients with Inclusion Body Myositis. A total of 9 subjects will be enrolled in the study. Subjects will be randomized to Part 1 or Part 2 of the study in blocks of 3 every 3 months.

Enrollment is anticipated to be staggered into 3 groups. The nine subjects will be randomized 2:1 in groups of 3 to early injections (Part 2) versus late (Part 1).

Stem cell injections will occur unilaterally in the flexor digitorum profundus muscles and the quadriceps group of muscles.

ELIGIBILITY:
Inclusion Criteria:

1. Meet any of the European Neuromuscular Centre Inclusion Body Myositis research diagnostic criteria 2011 categories for IBM. (see Appendix 3)
2. Demonstrate being able to arise from a chair without support from another person or device. Subjects may use their arms to push up.
3. Able to ambulate at least 20 ft/6 meters with or without assistive device. Once arisen from the chair, participant may use any walking device, i.e. walker/frame, cane, crutches, or braces. They cannot be supported by another person and cannot use furniture or wall for support.
4. Age at onset of weakness > 45 years
5. Able to give informed consent
6. Muscle strength graded between 6 and 9 for finger flexion and knee extension unilaterally on one side of the body (right or left) using the Kandell 0-10 scale. A subject may meet this criterion bilaterally and still be included in the study.

Exclusion Criteria:

1. History of any of the following excludes subject participation in the study: chronic infection particularly HIV or Hepatitis B or C; cancer other than basal cell cancer less than five years prior, or other chronic serious medical illnesses.
2. Presence of any of the following on routine blood screening: WBC < 3000; platelets < 100,000; hematocrit < 30%; BUN > 30 mg/dL; creatinine > 1.5 x upper limit of normal; symptomatic liver disease with serum albumin < 3 g/dl
3. History of most recent creatine kinase >15x the upper limit of normal without any other explanation besides IBM.
4. History of non-compliance with other therapies.
5. Use of testosterone except for physiologic replacement doses in case of androgen deficiency. Participants must have documented proof of the androgen deficiency.
6. Coexistence of any other neurological, cardiac, pulmonary, psychiatric, or rheumatologic disease that would likely to affect outcome measures.
7. Drug or alcohol abuse within past three months. Patient has recent history (within 6 months before Screening) of chronic alcohol or drug abuse which may compromise the patient's safety or ability to participate in study activities.
8. Use of cannabis
9. Participation in a recent drug study in the last 30 days prior to the screening visit or use of biologic agents less than 6 months prior to the screening visit.
10. Women who are lactating or pregnant, or men or women unwilling to use a highly effective method of birth control if not surgically sterile (defined as bilateral tubal ligation, bilateral oophorectomy, or hysterectomy for women; vasectomy for men) for both male and female participants until 4 weeks after last dose. Pre-menopausal women must have a negative pregnancy test prior to dosing with trial medication. Acceptable methods of birth control are:

    i. Hormonal methods associated with inhibition of ovulation such as oral, implantable, injectable, or transdermal contraceptives for a minimum of 1 full cycle (based on the patient's usual menstrual cycle period) before IMP administration.

    ii. Total abstinence from sexual intercourse since the last menses before IMP administration. (The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject. Periodic abstinence (calendar, symptothermal, post-ovulation methods), are not acceptable methods of contraception).

    iii. Intrauterine device (IUD) or intrauterine hormone-releasing system (IUS). If the subject is a sexually active male with female partners of child-bearing potential (postmenarchal)* he must use a condom with or without spermicide in addition to the birth control used by his partners during the trial until 3 months after the last dose of trial medication. *Non child-bearing potential is defined as post-menopausal (minimum of 12 months with no menses and follicle-stimulating hormone in the post-menopausal range) or sterilisation (hysterectomy, oophorectomy, or bilateral tubal ligation).
11. Participants taking corticosteroids within the previous 30 days prior to screening. Participants on intravenous immunoglobulin (IVIg) or other immunosuppressants within the last 3 months. Topical, nasal, and ocular corticosteroids are allowed unless they are being widely applied or the severity of the underlying condition makes them unsuitable in the Investigator's opinion. Local steroid injections are allowed.
12. Patients who have aPTT (Activated Partial Thromboplastin Time) values ≥ 1.8 X the normal value.
13. Patients who have received any anticoagulant within 1 hour prior to liposuction.
14. Patients who have received any anticoagulant within 1 hour of stem cell procedure
15. Patients who are on substantial anticoagulation (eg: GIIb/IIIa inhibitor class drugs) who cannot stop it within two weeks prior to adipose harvest
16. Participants who's IBM age of onset is under of 45
17. Participants with an elevated alkaline phosphatase level which may indicate Paget disease
18. Participants allergic or sensitive to lidocaine and or epinephrine
19. Participants with known drug exposures associated with neuromuscular side effects including antimalarial drugs (eg, chloroquine, hydroxychloroquine), colchicine, glucocorticoids, cholesterol-lowering drugs (eg, HMG-CoA reductase inhibitors [statins]) except if on stable dose for more than a year without impact on IBM progression, alcohol abuse, and cocaine
20. Use of other concomitant myositis treatment drugs, or cell or gene therapies (e.g. Arimoclomol, Bimagrumab, Follistatin, Rapamycin)
21. Any patient with an area of active skin infection at the site of lipoharvest
22. Participants that are current smokers, defined as an adult who has smoked 100 cigarettes in his or her lifetime and who currently smokes cigarettes.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
Safety (Frequency and Severity of Adverse Events) | 3 months post treatment
  The primary endpoint of safety will be reported as counts of subjects experiencing adverse events events (including abnormal laboratory results and vital signs). Six months after the first participant is treated, safety and efficacy will be accessed in order to make a decision about whether to continue the trial. Measures of safety will be reported for the last visit observed for each participant

SECONDARY OUTCOMES:
Change in Inclusion Body Myositis Functional Rating Scale (IBMFRS) from Baseline | 6 months post treatment
  The IBMFRS is a quickly administered (10-minute) ordinal rating scale used to determine participants' assessment of their capability and independence. It includes 10 measures (swallowing, handwriting, cutting food and handling utensils, fine motor tasks, dressing, hygiene, turning in bed and adjusting covers, changing position from sitting to standing, walking, and climbing stairs), graded on a Likert scale from 0 (being unable to perform) to 4 (normal). The sum of the 10 items gives a value between 0 and 40, with a higher score representing less functional limitation.
Change in Modified Timed Up and Go (mTUG) from Baseline | 6 months post treatment
  We will measure the patient's ability to get up from a chair allowing participants to use their arms (since most with sIBM cannot perform the task without pushing off), walk 3 meters, turn around and walk back to the chair and sit down. The use of nearby walls, or assistance from a caregiver is not allowed. This test will be performed twice and the fastest time will be used in the data analysis.
Change in Health Assessment Questionnaire-Disability Index (HAQ-DI) from Baseline | 6 months post treatment
  This is a self-report functional status measure based on the patient-centered dimension of disability.
Change in Patient Global Impression of Change from Baseline | 6 months post treatment
  The Patient Global Impression of Change (PGIC) is an assessment by the subject of self-perceived change in ability to conduct daily activities since the start of study medication. The scale ranges from 'very much worse' to 'much worse,' 'a little worse,' 'no change,' 'a little improved,' 'much improved,' and 'very much improved'.
Change in Manual Muscle Testing (MMT) from Baseline | 3, 6, and 12 months post treatment
  Manual muscle testing occurs when the evaluator records strength by having the subject resist while pushing on certain muscle groups with their arms and hands. MMT will include bilateral Knee Extension and Finger Flexion on the Kendall modification of the MRC scale being 0-10 scale.
Change in Handheld Dynamometry (HHD) from Baseline | 6 months post treatment
  HHD will be done using a MicroFET2 hand myometer. This is a hand-held device that allows the examiner to push against a muscle while the patient resists. Unlike the manual muscle test which provides a range, this device will provide an actual number. Knee extension will be tested bilaterally.
Change in Grip Strength from Baseline | 6 months post treatment
  Grip strength is done with the use of a Martin Vigorimeter that will measure grip strength. The maximum force generated by the patient from the two trials is used for each muscle group.

CONTACTS AND LOCATIONS:
Overall Officials: Mazen Dimachkie, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
During the conduct of the study, data about recruitment and data completeness will be shared with study personnel and appropriate regulatory and FDA oversight bodies. After completion of the study and analysis of the primary and secondary outcomes per protocol, a de-identified data set will be made available to any investigator interested in pursuing post-hoc analysis to aid in the overarching goal of bringing new therapies to IBM. Upon completion of the study data will be archived and listed with clinicaltrials.gov. In addition, data on process improvements will be made available to researchers interested in the innovations proposed in this study. KUMC will maintain a de-identified data set at completion which will be available to IBM researchers. We will ensure the results of the trial are widely distributed. At study completion we will announce the study in the The Myositis Association newsletter.
Supporting Information: SAP, CSR
Time Frame: Data should be available 6 months after the completion of the study and will be available indefinitely.